CLINICAL TRIAL: NCT06797024
Title: An Early Exploratory Clinical Study of the Safety, Tolerability, and Preliminary Efficacy of JY231 Injection for the Treatment of Relapsed/Refractory Neurologic Immune Disorders
Brief Title: JY231 Injection for the Treatment of Relapsed/Refractory Neurologic Immune Disorders
Acronym: JY231 NID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Daishi Tian, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-004
Record Dates: First submitted 2025-01-19; First posted 2025-01-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Diseases of the Nervous System
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY231 injection for the treatment of relapsed/refractory neurologic immune disorders (Experimental): JY231 Injection for the Treatment of relapsed/refractory neurologic immune disorders subjects who meet the inclusion criteria will receive intravenous JY231. JY231 infusion will produce CAR-T cells in the body.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — JY231 injection is administered intravenously and produces autologous CAR-T cells in the patient's body some time after infusion. A total of 3 dose groups were established to conduct a 3+3 dose-escalation study. The doses were divided into two categories: non-lymphodepletion and lymphodepletion pretreatment. The three dose groups for lymphodepletion included: 2×10^8 TU, 4×10^8 TU, and 8×10^8 TU. The three dose groups for non-lymphodepletion included: 2×10^9 TU, 4×10^9 TU, and 8×10^9 TU. The decision to perform lymphodepletion was based on the lymphocyte count and function during the patient screening period.

SUMMARY:
his study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed/refractory neurologic immune disorders. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed/refractory neurologic immune disorders.

DETAILED DESCRIPTION:
This open-label, single-arm study is designed to evaluate the efficacy and safety of in vivo CAR-T cell therapy in patients with relapsed/refractory neurologic immune disorders. Upon enrolment, leukapheresis will be performed and patients will receive 3-5 days of fludarabine and cyclophosphamide lymphodepleting therapy followed by an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be evaluated for safety and efficacy for up to 24 months to determine if the disease is under control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects (both 18 and 75 years of age) aged 18 to 75 years who have signed an informed consent (ICF) that none of the available treatment options have been effective; and
2. Previously diagnosed relapsed/refractory neuroimmune disorders for which there are currently no effective treatments, as determined by the specified diagnostic criteria, including:

Patients with AQP4 antibody-positive optic neuromyelitis optica (NMOSD) who meet the 2015 IPND NMOSD diagnostic criteria and meet one of the following requirements:

Treatment with at least one immunosuppressive agent for at least one year, or intolerance of immunosuppressive therapy with suboptimal symptom control; At least 2 relapses in the last 12 months or 3 relapses in the last 24 months and at least 1 relapse in the 12 months prior to screening.

Patients with myasthenia gravis (MG) who meet the 2020 MGFA diagnostic criteria for a total MG-ADL score of ≥6 with a relevant antibody-positive MGFA classification II-IV and meet one of the following requirements:

Have used standardized treatment with at least one immunosuppressive agent for more than 1 year and have one of the following poorly controlled conditions: 1) persistent weakness that interferes with daily life 2) exacerbation of MG symptoms and/or crisis episodes despite standardized treatment, and 3) inability to tolerate immunosuppressive therapy; Requires plasma exchange or intravenous gammaglobulin maintenance therapy.

Patients with chronic inflammatory demyelinating polyneuropathy (CIDP) who meet the 2021 EAN/PNS diagnostic criteria of an INCAT Disability Scale total score of 2-9 positive for relevant antibodies and meet one of the following requirements:

Standardized use of at least one first-line therapy for more than 3 months (cortisol hormone therapy, gammaglobulin, or plasma exchange therapy) with poor symptom control; Inability to tolerate cortisol hormone, gammaglobulin, and plasma exchange therapy because of side effects or other conditions.

Patients with a clinical diagnosis of refractory antibody-positive idiopathic inflammatory myopathy who meet the 2017 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for a diagnosis of IIM, with proximal muscle strength of at least one limb less than or equal to grade 4, and elevated creatine kinase. And meet one of the following requirements:

Presence of at least one creatine enzyme (CK, AST, ALT, ALD, LDH) ≥1.5 x ULN in the screening period; or dermatomyositis with a Dermatologic Lesion Extent and Severity Index (CDASI) ≥6; or evidence of active myositis in at least one of the following: MRI, electromyography, and muscle biopsy within the last 6 months; Presence of at least 1 myositis-specific (MSA), associated antibody (MAA), or antinuclear antibody (ANA) positive; Treatment with corticosteroids for at least 1 month and standardized treatment with at least one immunosuppressant/modulator (e.g., azathioprine, methotrexate, merti-macrolide, cyclosporine, tacrolimus, cyclophosphamide, leflunomide, and intravenous gammaglobulin) for more than 3 months with poor symptom control.

Inability to tolerate treatment with the above traditional regimens because of side effects or other conditions;

Clinically confirmed diagnosis of progressive MS (including primary progressive PPMS or secondary progressive SPMS) or relapsing-remitting RMS according to the 2017 Revised McDonald's Diagnostic Criteria; and Disability Status at Screening meets an EDSS score of 2-7, inclusive.RMS subjects will be required to standardize their use of DMT prior to signing the informed consent form medications still have a clear record of meeting the following conditions:

2 relapses documented within 2 years prior to screening, or

1 relapse documented within 1 year prior to screening, or Positive Gd-enhanced MRI scan within 1 year prior to screening (Screening MRI scan results may be used if no documented positive Gd-enhanced scan results existed in the previous year).

A clinically confirmed diagnosis of autoimmune encephalitis according to the 2016 International Autoimmune Encephalitis Diagnostic Criteria, along with all of the following requirements:

Positive test for at least one relevant autoantibody; Poor symptom control or intolerance of previous standardized treatment with glucocorticoids, at least one immunosuppressant/modulator including CD20 monoclonal antibody; Autoimmune encephalitis exacerbation within 3 months prior to signing the informed consent form; Disability status at screening meeting an mRS score of ≥2 or a CASE score of ≥4.

A clinically confirmed diagnosis of MOGAD according to the 2023 International Diagnostic Criteria for MOGAD, as well as meeting all of the following requirements:

Positive MOG autoantibody test by CBA method; Disability status at screening meeting an mRS score of ≥2; Poor symptom control or intolerance after prior standardized treatment with glucocorticoids, conventional immunosuppressants/modulators, and at least one biologic agent including CD20 monoclonal antibody.

3)ECOG 0 to 1 point; 4)Vital organ function assessment meets the following criteria: Blood: hemoglobin ≥ 60 g/L, platelet count ≥ 30 x 109/L; cardiac function: left ventricular ejection fraction (LVEF) ≥55%, ECG without obvious abnormalities; renal function: eGFR ≥30 ML/min/1.73m2; Liver function: AST and ALT ≤3.0 ULN, total bilirubin ≤2.0 ULN; Lung function: dlco ≥40% of predicted value; fvc ≥50% of predicted value; have criteria for single or venous blood collection and no other contraindications to cell collection; 5)Subjects of childbearing age with negative urine pregnancy test results and agree to use effective contraception for the duration of the trial until 1 year post-infusion; 6)The patient or his/her guardian agrees to participate in the clinical trial and signs the informed consent form, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. have a contraindication or hypersensitivity to fludarabine, cyclophosphamide, and any component of the test drug;
2. have received intravenous immunoglobulin or plasma exchange therapy or immunosorbent therapy within 4 weeks prior to retrieval;
3. have used tacrolimus, cyclosporine, azathioprine, morphimecrolimus, mycophenolate mofetil, methotrexate, or methotrexate within 1 week prior to mono-harvesting;
4. Treatment with neonatal Fc receptor (FcRn) antagonists (e.g., Efgartigimod, etc.) within 1 week prior to single-take;
5. have used complement inhibitory therapy (e.g., eculizumab, etc.) within 1 week prior to single-take;
6. Suffering from severe cardiac, hepatic, pulmonary, hematologic, or endocrine system diseases that, in the judgment of the investigator, pose a greater risk than benefit of participation in the trial;
7. Presence of active or uncontrollable infection requiring systemic therapy within 1 week prior to screening;
8. Previous hematopoietic stem cell transplantation or solid organ transplantation (except cornea and hair transplantation), or Grade 2 or higher acute graft-versus-host disease (GVHD) within 2 weeks prior to screening;
9. Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) positive and peripheral blood Hepatitis B Virus (HBV) DNA titer test is greater than the normal reference value range; or Hepatitis C Virus (HCV) antibody positive and peripheral blood Hepatitis C Virus (HCV) RNA titer test is greater than the normal reference value range; or Human Immunodeficiency Virus (HIV) antibody positive; or positive syphilis test; or positive cytomegalovirus (CMV) DNA test;
10. Have received a live vaccine within 4 weeks prior to screening;
11. Positive pregnancy test;
12. Patients with malignant diseases such as malignant tumors prior to screening, except adequately treated carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
13. Patients who have participated in another clinical trial within 3 months prior to screening;
14. Other conditions that the investigator considers unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dai-shi Tian, PhD, Principal Investigator — Tongji Hospital; Wei Wang, PhD, Principal Investigator — Tongji Hospital; Chuan Qin, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No